CLINICAL TRIAL: NCT01442077
Title: Low Intensity Extracorporeal Shock Wave Therapy for the Treatment of Erectile Dysfunction- 4 Arms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0359-11-RMB
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- arm 1 (Active Comparator): Series of 12 treatments, in which the subject will be treated twice a week for 3 weeks (6 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for 3 weeks (6 treatments.
  Interventions: Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000)
- arm 2 (Active Comparator): Series of 12 treatments, in which the subject will be treated twice a week for 6 consecutive weeks, without intermission.
  Interventions: Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000)
- arm 3 (Active Comparator): Series of 8 treatments, in which the subject will be treated twice a week for two weeks (4 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for two weeks (4 treatments).
  Interventions: Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000)
- arm 4 (Active Comparator): Series of 6 treatments, in which the subject will be treated once a week for 3 weeks (3 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated once a week for 3 weeks (3 treatments).
  Interventions: Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000)

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000) — Series of 12 treatments, in which the subject will be treated twice a week for 3 weeks (6 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for 3 weeks (6 treatments).
  Other Names: No other names
Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000) — Series of 12 treatments, in which the subject will be treated twice a week for 6 consecutive weeks, without intermission.
  Other Names: No other names
  Arms: arm 2
Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000) — Series of 8 treatments, in which the subject will be treated twice a week for two weeks (4 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for two weeks (4 treatments).
  Other Names: No other names
  Arms: arm 3
Device: Extracorporeal Shockwave Therapy Generator (Omnispec ED1000) — Series of 6 treatments, in which the subject will be treated once a week for 3 weeks (3 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated once a week for 3 weeks (3 treatments).
  Other Names: No other names
  Arms: arm 4

SUMMARY:
Low intensity shock waves(LISW) have been proven in animal studies to induce local growth of new blood vessels. The investigators hypothesized that LISW therapy could improve the symptoms of patients with erectile dysfunction resulting from a problem of blood supply who respond to oral therapy (PDE-5 inhibitors). The current study will check 4 different arm.

DETAILED DESCRIPTION:
At the first meeting the patient will receive a full explanation of the study, the potential efficacy and risks. After that the patient will be asked to sign an informed consent form, and will be asked about general medical condition and any problems related to sexual dysfunction. Than the patient's sexual function will be assessed by sexual function questionnaires. The criteria for inclusion and exclusion will be reviewed, as well as physical examination. During the visit, the patient will be assigned to one arm of the study (random), and by the arm he belongs he will receive an explanation about this procedure. Then shall obtain reporting sexual encounter diaries (SEP) and will be asked to avoid using PDE5i's for a month (washout), then it would be the first visit. At the first visit (Visit 1) The patient will be questioning the sexual function questionnaires without PDE5i's and will pass examination performance Endothelial - FMD, the test takes about 10 minutes, it is not an invasive test (not involved in inserting an instrument or any medication) and is painless. The patient may be asked to also undergo Doppler ultrasound. At the end of the visit 1 the patient will begin treatment series and will continue to study under the arm belongs, as described: 1.Series of 12 treatments, in which the subject will be treated twice a week for 3 weeks (6 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for 3 weeks (6 treatments). 2.Series of 12 treatments, in which the subject will be treated twice a week for 6 consecutive weeks, without intermission. 3.Series of 8 treatments, in which the subject will be treated twice a week for two weeks (4 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated twice a week for two weeks (4 treatments). 4.Series of 6 treatments, in which the subject will be treated once a week for 3 weeks (3 treatments), then would be discontinuation of the study for 3 weeks, and at the end of this period will be treated once a week for 3 weeks (3 treatments).

Four weeks after the treatment series ends the patient will come for another visit will be asked to fill in questionnaires and perform the FMD test again.

ELIGIBILITY:
Inclusion Criteria:

* ED for more than six months in duration.
* At least 50% unsuccessful sexual intercourses for 4 attempts at 4 different days.
* Previous positive experience with PDE5iswithin the past six months.
* A minimum of two sexual attempts per month.
* An IIEF-ED domain score of ≥19, post screening PDE5i intake.
* An IIEF-ED domain score of ≥17 and a Rigidity score ≥ 3 , post screening with PDE5i intake
* A Rigidity score ≥ 3 post screening PDE5i intake.
* A stable heterosexual relationship with the same partner for more than three months.
* Delta IIEF-ED domain score ≤5 points on visit 1 (after 1 month wash out) compared to the IIEF-ED domain score on screening.

Exclusion Criteria:

* Prior prostate surgery.
* Any cause of ED other than of vascular etiology.
* Any unstable medical or psychiatric condition, spinal cord injury, or penile anatomical abnormalities including Peyrone's disease.
* Clinically significant chronic hematological disease.
* Cardiovascular conditions that prevent sexual activity.
* History of heart attack, stroke, or life-threatening arrhythmia within 6 months prior to enrollment into the study.
* Cancer within the past five years.
* Use of anti-androgens, or oral or injectable androgens
* Use of any other treatments for ED that includes oral medications, vacuum devices, constrictive devices, injections, or urethral suppositories within seven days of screening.
* Hormonal, neurologic, or psychological pathology.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Increase in IIEF ED Domain Questionaire of >5 is considered as a treatment success | 3 months

SECONDARY OUTCOMES:
Rigidity Score Questionaire- an increase of at least 1 point is considered as a treatment success | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel